CLINICAL TRIAL: NCT01865253
Title: Renal Denervation for Complicated Hypertension (RDNP-2012-03)
Brief Title: Renal Denervation for Complicated Hypertension
Acronym: RDNP-2012-03
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No new participants enrolled. Protocol superseded.
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 087/12; 1034397 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Hypertension
Keywords: renal denervation; blood pressure; cardiovascular risk; target organ damage; sympathetic activity; chronic kidney disease; non-compliance
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation (Experimental): Renal Denervation treatment
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — Renal Denervation
  Other Names: Symplicity Renal Denervation Catheter

SUMMARY:
This is an observational proof of concept study investigating the safety and effectiveness of renal denervation to lower blood pressure in people whose blood pressure is not adequately controlled due to:

* intolerance to antihypertensive medication
* inability to take antihypertensive medication due to planned pregnancy
* renal artery stenosis
* chronic kidney disease
* non-compliance to antihypertensive medication

A total of 125 participants, 25 from each of the groups mentioned above will be recruited to the study.

The duration of this study is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* BP ≥140/90 mmHg (or ≥130/80 mmHg for patients with diabetes)
* Intolerance to ≥2 antihypertensive drug classes
* Inability to take Angiotensin-Converting-Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blockers (ARBs) or Direct Renin inhibitors (DRIs) due to planned pregnancy
* Renal artery stenosis
* Chronic Kidney Disease

Exclusion Criteria:

* renal artery anatomy ineligible for treatment
* individual has had myocardial infarction, unstable angina or cerebrovascular accident within 6 months of screening visit
* female participants of childbearing potential must have negative pregnancy test prior to treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in average office blood pressure | baseline to 6 months post procedure
  Change in systolic and diastolic average office blood pressure from baseline to 6 months post procedure

SECONDARY OUTCOMES:
Blood pressure control | baseline to 6 months post procedure
  Percentage of patients who achieved BP target at 6 months post procedure
Number of drugs required to reach target blood pressure | baseline to 6 months post procedure
  Number of drugs required to reach target blood pressure
Time to achieve blood pressure target | baseline to 6 months post procedure
  Time to achieve blood pressure target
Change in sympathetic nerve activity | baseline to 6 months post procedure
  Change in muscle sympathetic nerve activity, renal and whole body Noradrenaline (NA) spillover
Change in left ventricular structure and function | baseline to 6 months post procedure
  Change in left Ventricular mass index, Ejection Fraction, diastolic filling
Change in Quality of life | baseline to 6 months post procedure
  Change in Quality of life as assessed by relevant questionnaires
Change in serum and urine Biochemistry | baseline to 6 months post procedure
  Plasma renin activity, aldosterone, estimated Glomerular Filtration Rate(eGFR), Urinary Albumin Creatinine Ratio (UACR), inflammatory markers, 24hour urine creatinine clearance, sodium, fasting glucose, fasting insulin, c peptide, Homeostasis Model Assessment (HOMA) index, lipid profile.
Change in markers of arterial stiffness | baseline to 6 months
  Change in markers of arterial stiffness including Augmentation Index (AI) and Pulse Wave Velocity (PWV)

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, MD, Principal Investigator — Baker IDI Heart & Diabetes Institute
Locations (1):
- Baker IDI Heart & Diabetes Institute, Melbourne, Victoria, Australia